CLINICAL TRIAL: NCT01741389
Title: The Role of Melatonin in the Regulation of Blood Coagulation
Acronym: COME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Sunnaas Hospital (Unknown); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2009/295
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injured, Tetraplegia
Keywords: Circadian variation, hemostasis, melatonin, tetraplegia
MeSH Terms: conditions — Quadriplegia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep only (Placebo Comparator): Placebo given at night to tetraplegic individuals before going to sleep,
  Interventions: Drug: Melatonin ("Circadin")
- Melatonin (Active Comparator): Melatonin given at night to tetraplegic individuals before going to sleep.
  Interventions: Drug: Melatonin ("Circadin")

INTERVENTIONS:
Drug: Melatonin ("Circadin")

SUMMARY:
The main aim is to examine the influence of daylight and melatonin on the temporal variations of hemostatic factors with key roles in the hemostatic process and its regulation. Particular emphasis will be on exploring the role of melatonin in hemostasis by comparing subjects with tetraplegia with able-bodied control subjects.

ELIGIBILITY:
Inclusion Criteria:

Intervention group:

* A diagnosis of tetraplegia for at least 2 years, and otherwise healthy.
* Must not use drugs permanently (except anti-spasmolytics).
* Must be able to swallow tablets.
* Must give written consent to participate.

Control group:

* Must be healthy.
* Must not use drugs permanently.
* Must give written consent to participate.

Exclusion Criteria:

Both groups:

* Those with acute or chronic co-morbidity.
* Unable to cooperate.
* Not provided written consent to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Circadian variation of hemostatic factors | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnaas Hospital, Nesodden, Nesodden, Norway

REFERENCES:
- [Background] Dahm A, Osterud B, Hjeltnes N, Sandset PM, Iversen PO. Opposite circadian rhythms in melatonin and tissue factor pathway inhibitor type 1: does daylight affect coagulation? J Thromb Haemost. 2006 Aug;4(8):1840-2. doi: 10.1111/j.1538-7836.2006.02048.x. No abstract available. PMID 16879232
- [Background] Kostovski E, Dahm AE, Iversen N, Hjeltnes N, Osterud B, Sandset PM, Iversen PO. Melatonin stimulates release of tissue factor pathway inhibitor from the vascular endothelium. Blood Coagul Fibrinolysis. 2011 Jun;22(4):254-9. doi: 10.1097/MBC.0b013e3283442ce2. PMID 21297449
- [Background] Dahm AE, Iversen PO, Hjeltnes N, Sandset PM. Differences in circadian variations of tissue factor pathway inhibitor type 1 between able-bodied and spinal cord injured. Thromb Res. 2006;118(2):281-7. doi: 10.1016/j.thromres.2005.07.021. Epub 2005 Aug 31. PMID 16139333